CLINICAL TRIAL: NCT02280772
Title: Effect of Glucomannan Supplementation on Body Weight in Overweight and Obese Children: A Randomized Controlled Trial
Brief Title: Effect of Glucomannan Supplementation on Body Weight in Overweight and Obese Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-2014
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Overweight
Keywords: glucomannan; obesity; children; overweight; adolescents; treatment
MeSH Terms: conditions — Obesity; Overweight | interventions — (1-6)-alpha-glucomannan; Amorphophallus konjac root extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucomannan (Experimental): Glucomannan orally, 3g/day (in three divided doses), for 12 weeks
  Interventions: Dietary Supplement: Glucomannan
- Maltodextrin (Placebo Comparator): Maltodextrin orally, 3g/day (in three divided doses), for 12 weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Glucomannan
  Other Names: Amorphophallus konjac
  Arms: Glucomannan
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
Glucomannan (GNN), a water-soluble dietary fiber derived from the plant Amorphophallus konjac, is marketed for weight reduction. The exact mechanisms by which GNN might exert its actions are unclear. Nonetheless, it has been shown that GNN slows gastric emptying by forming a viscous gel of large volume, which increases the feeling of satiety. Current evidence on the effectiveness of GNN for weight reduction is sparse, and well-designed trials performed in children are needed to assess the efficacy of this modality. We aim to systematically evaluate the efficacy of GNN consumption for the management of overweight and obesity in children.

DETAILED DESCRIPTION:
Methods and analysis

Children aged 6 to 17 years with overweight and obesity (based on the WHO growth criteria) will be randomly assigned to receive GNN or placebo (maltodextrin) (both at a dose of 3 g/day) for 3 months and will be followed up for 3 months. Prior to the intervention, all children will receive dietetic advice, and they will be encouraged to engage in physical activity. The primary outcome measure will be the BMI-for-age z-score difference between the groups at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 6-17 years;
* overweight or obesity based on the WHO (World Health Organization) growth charts/references (>+1 standard deviation [SD] or >+2 SD, respectively)

Exclusion Criteria:

* drug therapy for a chronic disease (including drugs that influence appetite or body weight);
* type 1 or 2 diabetes;
* history of surgical treatment of obesity;
* participation in another program for treating obesity during the project and/or 3 months prior to recruitment;
* secondary causes of obesity;
* pregnancy.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
BMI-for-age z-score difference | 0-12 weeks
  Baseline versus end of the intervention

SECONDARY OUTCOMES:
Body composition | 0-13 weeks
  Whole body fat, central body fat, fat-free mass (grams) assessed by a dual energy X-ray absorption (DXA)
BMI-for-age z-score difference | 0-24 weeks
  Baseline versus end of the follow-up
Proportion of participants with dyslipidemia | At baseline, 12 weeks and 24 weeks
  Proportion of participants with dyslipidemia from baseline to week 12 and week 24 (mean change, SD)
Proportion of participants with impaired fasting plasma glucose (FPG) | At baseline, 12 weeks and 24 weeks
  Proportion of participants with impaired fasting plasma glucose (FPG) from baseline to week 12 and week 24 (mean change, SD).
Energy intake (kJ/d) | At baseline and at week 12, week 24.
  Based on self-written, 3-day food records
Physical activity | at baseline and at week 12
  Measured using an accelerometer
Adverse events | 0-12 weeks
Blood pressure (systolic and diastolic) | Baseline, week 12, 24 weeks.
  The mean change from baseline to week 12, and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bartlomiej M Zalewski, MD, Principal Investigator — The Medical University of Warsaw; Hanna Szajewska, Professor, Study Chair — The Medical University of Warsaw
Locations (1):
- The Medical University of Warsaw, Department of Paediatrics, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Derived] Zalewski BM, Szajewska H. No Effect of Glucomannan on Body Weight Reduction in Children and Adolescents with Overweight and Obesity: A Randomized Controlled Trial. J Pediatr. 2019 Aug;211:85-91.e1. doi: 10.1016/j.jpeds.2019.03.044. Epub 2019 Apr 26. PMID 31036412
- [Derived] Zalewski BM, Szajewska H. Effect of glucomannan supplementation on body weight in overweight and obese children: protocol of a randomised controlled trial. BMJ Open. 2015 Apr 13;5(4):e007244. doi: 10.1136/bmjopen-2014-007244. PMID 25869689